CLINICAL TRIAL: NCT06520280
Title: Comparative Study Between Injection Molding and Additive Manufacturing Complete Denture Bases Construction Techniques: an in Vivo Study
Brief Title: Comparative Study Between Injection Molding and Additive Manufacturing Complete Denture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ibrahim Mohamed Ali Ibrahim Abd Elrahman (Other)
Responsible Party: Sponsor-Investigator, Ibrahim Mohamed Ali Ibrahim Abd Elrahman, prosthodontist, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 875/281
Record Dates: First submitted 2024-07-21; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Complete Denture
MeSH Terms: interventions — Nylons

STUDY DESIGN:
Intervention Model Description: Group I: First, patients will receive maxillary and mandibular complete dentures constructed by polyamide thermoplastic resin. Group II: First, patients will receive maxillary and mandibular complete dentures constructed by 3D printed
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GroupI (Other): First, patients will receive maxillary and mandibular complete dentures constructed by polyamide thermoplastic resin.
  Interventions: Other: polyamide and 3D printed complete denture
- Group II (Other): First, patients will receive maxillary and mandibular complete dentures constructed by 3D printed
  Interventions: Other: polyamide and 3D printed complete denture

INTERVENTIONS:
Other: polyamide and 3D printed complete denture — pts. receive 2 sets of complete dentures made from polyamide and 3d printed to use

SUMMARY:
The objective of the trial is to compare between of polyamide and rapidly prototyped (3D-printed) complete denture bases regarding retention, patient satisfaction, masticatory efficiency and microbial adhesion.

DETAILED DESCRIPTION:
completely edentulous male patients will be selected from the out patient clinic of Removable Prosthodontic Department, Faculty of Oral and Dental medicine Al-Azhar University (Boys), Cairo, Egypt. patients will be selected and divided into randomly two equal groups and each patient will receive two sets of complete dentures: Group I: First, patients will receive maxillary and mandibular complete dentures constructed by polyamide thermoplastic resin. Group II: First, patients will receive maxillary and mandibular complete dentures constructed by 3D printed. Retention will be measured for all patients at delivery day, one month after delivery and three months after delivery. After that, there will be 2 weeks as a period of rest and the two groups will be reversed with reassessment at the same time interval. Patient satisfaction will be measured for all patients after 1 and 3 months follow up through a validated questionnaire. Masticatory efficiency will be measured by measuring muscle activity of the masseter and anterior fibers of the temporalis muscle on both sides for both dentures at one week, one month and three months after delivery using electromyography with three types of test foods. Microbial adhesion Samples will be collected one month after delivery of dentures, swaps will be taken from the fitting palatal surface of the upper denture, this will be done immediately after removal of the denture.

ELIGIBILITY:
Inclusion Criteria:

1. Completely edentulous male patients ranging from age 45 to 60 years.
2. Angle's Class I skeletal relationship.
3. Well-developed ridge with U-shaped palatal vault and adequate firm mucosa.
4. Last extraction took place six months ago.
5. Normal facial symmetry.
6. Cooperative patients.

Exclusion Criteria:

1. Temporomandibular disorders.
2. Uncontrolled diabetes.
3. Flabby tissues or sharp mandibular residual ridge.
4. Smokers.
5. Patients with neuromuscular disorders.
6. Patients on chemotherapy or radiotherapy.
7. Severe psychiatric disorders.
8. Angle's class II and III skeletal relationship

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
retention | 6 months
  Retention will be measured for all patients at delivery day, one month after delivery and three months after delivery. After that, there will be 2 weeks as a period of rest and the two groups will be reversed with reassessment at the same time interval.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed helal, professor, Study Director — AZU
Locations (1):
- Faculty of Dental Medicine, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: comparison of retention between maxillary milled and conventional denture bases: A clinical study. — https://pubmed.ncbi.nlm.nih.gov/27765399/
- See also: Accuracy and retention of denture base fabricated by heat curing and additive manufacturing. — https://pubmed.ncbi.nlm.nih.gov/30584053/
- See also: Comparison between Retention of Maxillary Acrylic and Nylon Denture Base Materials. — https://polytechnic-journal.epu.edu.iq/home/vol10/iss1/7/